CLINICAL TRIAL: NCT04746521
Title: DEtection of Cellular-MEdiated immuniTy in COVID-19 Patients and Subjects Who undeRgone vAccination Program
Brief Title: Cellular-Mediated Immunity in COVID-19
Acronym: DEMETRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: L. Vanvitelli
Record Dates: First submitted 2021-02-08; First posted 2021-02-09 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Thromboembolism
MeSH Terms: conditions — COVID-19; Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood, genomic DNA, RNA, and proteins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Severe COVID-19 hospitalized patients: A total of 50 severe COVID-19 patients admitted to the Sub-Intensive Care Unit of A.O.R.N. Ospedali dei Colli, Cotugno Hospital, Naples (Italy) will be recruited, of which N=50 with thromboembolic complications (PE+) and N=50 without thromboembolic complications (PE-) balanced for age and sex of individuals.
  Interventions: Biological: genomicDNA extraction
- Healthy controls (comparator group): As control group (CTRL), we will recruit a total of N=50 healthy subjects (never diagnosed with Sars-Cov2 infection) among the volunteer blood donors attending the U.O.C. Divisione di Immunologia Clinica, Immunoematologia, Medicina Trasfusionale e Immunologia dei Trapianti, Dipartimento di Medicina Interna e Specialistica, AOU, "L. Vanvitelli" University of Campania (Naples, Italy).
  Interventions: Biological: genomicDNA extraction
- COVID-19 patients compared with vaccinated subjects: 1. Patients with previous Sars-CoV-2 infection who did not undergo vaccination;
  2. Patients with previous Sars-CoV-2 infection who undergone vaccination
  3. Subjects without previous Sars-CoV-2 infection who undergone vaccination
  Interventions: Diagnostic Test: Multitest 6 color TBNK and BD Lyotubes

INTERVENTIONS:
Diagnostic Test: Multitest 6 color TBNK and BD Lyotubes — The Multitest 6 color TBNK allows us to count the population-specific B, T, NK cells
  Groups: COVID-19 patients compared with vaccinated subjects
Biological: genomicDNA extraction — Peripheral blood biospecimens (about 10-15 mL) will be collected through venipuncture in EDTA tubes. Peripheral blood mononuclear cells (PBMCs) will be isolated using Ficoll® Paque Plus (Sigma-Aldrich) centrifugation gradient and genomic DNA will be extracted from fresh PBMCs using DNeasy Blood & Tissue kit (QIAGEN), according to manufacturer protocols
  Groups: Healthy controls (comparator group); Severe COVID-19 hospitalized patients

SUMMARY:
In order to prevent reinfection, it is needed to detect the cellular-mediated immune response to the Sars-CoV-2 infection. The first goal of this study will be to detect the cellular-mediated immune response in patients affected by COVID-19 (with or without vaccination) and healthy subjects who undergone vaccination program. The second goal of this study will be to identify the genetic and epigenetic biomarkers that influence individual immunological response and clinical evolution to the severe manifestations of the COVID-19.

DETAILED DESCRIPTION:
First goal: Characterization of the immune response using detailed phenotypic evaluation of the adaptive compartment comprising B, T, and NK cells. The Investigators aim is to detect the cellular-mediated immune response in patients affected by COVID-19 and subjects who undergone vaccination program.

The Investigators will recruit three classes of subjects:

1. Patients with previous Sars-CoV-2 infection who did not undergo vaccination;
2. Patients with previous Sars-CoV-2 infection who undergone vaccination;
3. Subjects without previous Sars-CoV-2 infection who undergone vaccination.

Second goal: Evaluation of genetic and epigenetic biomarkers that influence individual immunological response and susceptibility to thromboembolic manifestations in severe COVID-19 hospitalized patients.

The Investigators will recruit:

1. A total of 50 severe COVID-19 patients admitted to the Sub-Intensive Care Unit of A.O.R.N. Ospedali dei Colli, Cotugno Hospital, Naples (Italy) of which N=50 with thromboembolic complications (PE+) and N=50 without thromboembolic complications (PE-);
2. A total of N=50 healthy subjects (never diagnosed with Sars-Cov2 infection) among the volunteer blood donors attending the U.O.C. Divisione di Immunologia Clinica, Immunoematologia, Medicina Trasfusionale e Immunologia dei Trapianti, Dipartimento di Medicina Interna e Specialistica, AOU, "L. Vanvitelli" University of Campania (Naples, Italy)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Previous diagnosis of COVID-19
* Absence of COVID-19 diagnosis

Exclusion Criteria:

* Age <18 years
* Inflammatory diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases:
  Patients with previous diagnosed Sars-CoV-2 infection who did undergo vaccination.
  Patients with previous diagnosed Sars-CoV-2 infection who did not undergo vaccination.
  Subjects without diagnosed Sars-CoV-2 infection who adhered to vaccination program.
  -
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-12-14 (Estimated)

PRIMARY OUTCOMES:
Detection of Cellular-Mediated Immune Response | 3 Months
  The Investigators will perform the BD Multitest 6-color TBNK by using 50 uL of peripheral blood to detect the absolute number (N) of CD3+, CD19+, CD16+, CD46+, CD4+ and CD8+ cells.
Detection of Cellular-Mediated Immune Response | 3 Months
  The Investigators will perform the BD™ Lyotubes kit by using 150 uL of peripheral blood to detect the absolute number (N) of CD4+ and CD8+ cells undergoing to differentiation from naive T cells to central memory, effector memory, and terminal memory

SECONDARY OUTCOMES:
Detection of T cell subpopulation maturation | 5 months
  The Investigators will perform the BD™ Lyotubes kit by using 150 uL of peripheral blood to detect the absolute number (N) of CD4+ and CD8+ cells undergoing to differentiation from naive T cells to central memory, effector memory, and terminal memory.
Detection of T cell subpopulation maturation | 5 months
  The Investigators will perform the BD™ Lyotubes kit by using 150 uL of peripheral blood to detect the % of CD4+ and CD8+ cells undergoing to differentiation from naive T cells to central memory, effector memory, and terminal memory.

CONTACTS AND LOCATIONS:
Locations (1):
- U.O.C. Division of Clinical Immunology, Immunohematology, Transfusion Medicine and Transplant Immunology, Regional Reference Laboratory of Transplant Immunology, Department of Internal and Specialty Medicine, A.O.U., UniversityofCampania "Luigi Vanvitelli, Napoli, Italy